CLINICAL TRIAL: NCT04074603
Title: Comparing the Effects of Insulin Glargine on Peripheral Blood Glucose Between Needle-free Jet Injection and Conventional Insulin Pen
Brief Title: Comparing the Effects of Insulin Glargine on Blood Glucose Between Needle-free Jet Injection and Insulin Pen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-hua Ma (Other)
Responsible Party: Sponsor-Investigator, Jian-hua Ma, Director, Head of Endocrinology department, Clinical Professor, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KY20190530-02-KS-01
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes
Keywords: Needle-free jet injection; Insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): needle-free before needle
  Interventions: Device: The needle-free jet injector
- Group B (Experimental): needlebefore needle-free
  Interventions: Device: Conventional insulin pen

INTERVENTIONS:
Device: The needle-free jet injector — Continuous insulin therapy for 2 weeks
  Arms: Group A
Device: Conventional insulin pen — Continuous insulin therapy for 2 weeks
  Arms: Group B

SUMMARY:
To comparing the blood sugar improvement and patient sensibility of insulin glargine injected with needle-free jet injector and conventional insulin pen

DETAILED DESCRIPTION:
Compared with conventional pen, needle-free jet injection of insulin has faster flow rate and larger area of local subcutaneous absorption. The aim of this study was to investigate the effects of subcutaneous insulin glargine injection with needle-free jet injection and conventional pen on blood glucose profile and safety in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and be able to sign informed consent prior to the trial.
* patients with type 2 diabetes, aged 18-80 years old, meeting WHO1999 diagnostic criteria, have not used any hypoglycemic drugs. The dosage of insulin glargine (4-35 units) combined with oral medicationis, stable for more than 2 months.
* No acute complications such as diabetic ketoacidosis, diabetic hyperosmolar syndrome, etc.
* Subjects are able and willing to monitor peripheral blood sugar and regularity of diet and exercise.

Exclusion Criteria:

* Patients with insulin allergy.
* Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value;Serum creatinine was 1.3 times higher than the upper limit of normal.
* Drug abuse and alcohol dependence in the past 5 years.
* Systemic hormone therapy was used in the last three months.
* Patients with poor compliance and irregular diet and exercise.
* Patients with pregnancy, lactation or pregnancy intention.
* Any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose changes | 2 weeks
  The effect of Needle-free Jet Injection and Insulin Pen injection Insulin Glargine on blood glucose changes in T2Dm
The glucose fluctuation | 2 weeks
  The effect of Needle-free Jet Injection and Insulin Pen injection Insulin Glargine on glucose profile (MAGE, 24h-MG, CV%, SDBG, TAR, TIR, TBR) changes in type 2 diabetes mellitus by FGM.

SECONDARY OUTCOMES:
Assessment of safety and tolerance | 2 weeks
  The effect of Needle-free Jet Injection and Insulin Pen injection Insulin Glargine on safety and tolerance changes in type 2 diabetes mellitus by Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided